CLINICAL TRIAL: NCT00309530
Title: A Prospectively Randomized Phase III Study on Adjuvant Chemotherapy and Adjuvant Chemo-Immunotherapy in Patients With Operated Colon Carcinoma Dukes C (Stage III; T1-4, N1-30, M0).
Brief Title: Randomized Study on Adjuvant Chemotherapy and Adjuvant Chemo-Immunotherapy in Colon Carcinoma Dukes C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG 90
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 1999-04

CONDITIONS: Colon Cancer Stage III
Keywords: Fluorouracil; Levamisol; Interferon; Colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Fluorouracil; Levamisole; Interferons

INTERVENTIONS:
Drug: 5-fluorouracil, levamisol, interferon

SUMMARY:
This clinical investigation examined the effectivity 5-fluorouracil, of adding levamisol or interferon to 5-fluorouracil, and of a 5-fluorouracil/levamisol/interferon triple combination, in terms of recurrence-free and overall survival in curatively operable colon carcinoma Stage III.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically verified, curatively operated colon carcinoma Stage III (R0, T1-4, N1-3, M0)
* Age: less than 80 years
* WHO Performace Status > 2
* Adequate bone marrow reserve
* Informed consent

Exclusion Criteria:

* Rectal cancer
* R1, R2, carcinosis peritonei
* Start of chemo- or chemo-immunotherapy > 42 days postop; other adjuvant radiotherapy, chemotherapy or immunotherapy
* Serious concomitant disease, in particular chronically inflammatory large intestine, cardiopathic disease, malignant second carcinoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598
Dates: Start 1990-10

PRIMARY OUTCOMES:
Recurrence-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Jakesz, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group
Locations (16):
- Austria (16):
  - Hospital Guessing, Güssing, Burgenland
  - Hospital Oberpullendorf, Oberpullendorf, Burgenland
  - Hospital BHB St. Veit/Glan, Surgery, Saint Veit A. D. Glan, Carinthia
  - State Hospital Wolfsberg, Wolfsberg, Carinthia
  - Paracelsus Medical University Salzburg - Oncology, Salzburg, Salzburg
  - Medical University of Graz, Oncology, Graz, Styria
  - State Hospital Leoben, Surgery, Leoben, Styria
  - Hospital St. Vinzenz, Zams, Tyrol
  - State Hospital Kirchdorf, Kirchdorf, Upper Austria
  - General Hospital Linz, Linz, Upper Austria
  - Hospital BHB Linz, Linz, Upper Austria
  - State Hospital Voecklabruck, Internal Medicine, Vöcklabruck, Upper Austria
  - Hospital Kreuzschwestern Wels, Wels, Upper Austria
  - Medical University Vienna, General Hospital, Vienna, Vienna
  - Wilheminenspital, Internal Medicin I, Vienna, Vienna
  - State Hospital Feldkirch, Feldkirch, Vorarlberg

REFERENCES:
- See also: Related Info — http://www.abcsg.at